CLINICAL TRIAL: NCT03643614
Title: Evaluation of Effectiveness and Safety of Autologous Adipose-derived Regenerative Cells Injection for Treatment of Radiation-induced Rectovaginal Fistula
Brief Title: Autologous Adipose-derived Regenerative Cells Injection for Treatment of Radiation-induced Rectovaginal Fistula
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: South Ural State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU SUSMU 310855.210617.1
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Rectovaginal Fistula
Keywords: adipose derived stromal cells; stromal vascular fraction; mesenchymal stem cells; rectovaginal fistula
MeSH Terms: conditions — Rectovaginal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Injection of autologous regenerative cells of adipose tissue for treatment of radiation induced rectovaginal fistulas
  Interventions: Procedure: Injection of autologous regenerative cells of adipose tissue

INTERVENTIONS:
Procedure: Injection of autologous regenerative cells of adipose tissue — Autologous regenerative cells of adipose tissue obtained by enzymatic digestion of lipoaspirate are injected diffusively in the submucosal plane of the rectum and vagina with a sharp 27G needle. Adipose tissue that has not been subjected to enzymatic processing is injected through the punctures on the skin into the deep layers of the rectovaginal septum by means of cannula of 1.0-1.2 mm in diameter, 70 mm in length, 0.1-0.2 ml in one retrograde pass of the cannula.

SUMMARY:
A new strategy for treatment of late radiation damage is to develop methods aimed at stimulating the regenerative capabilities of irradiated tissues. Since the main pathogenetic mechanism of the development of late radiation damage is the death or damage of the replicative mechanism of stromal cells (SC), a justified approach can be considered as transplantation of intact SC. Currently, there is convincing evidence in the scientific literature that the injection of intact autologous SCs into the zone of fibrosis surrounding the chronic radiation ulcer leads to the healing of a wound defect.

An Initiative Clinical Trial. Introduction of autologous regenerative cells of adipose tissue for the treatment of post-irradiation vaginal-rectal fistula. It is assumed that patients will be included in the project within 12 months; the monitoring of each patient will last for 6 months; the total duration of the clinical part of the study will be 18 months; The total duration of the clinical trial including the preparatory phase and the writing of the report is about 24 months. It is assumed that at least 16 patients aged 20 to 75 years who have verified diagnosis of post-irradiation vaginal-rectal fistula will participate in this pilot project. The aims of the clinical trial are to preliminarily assess the safety, effectiveness and quality of life of patients after introducing autologous regenerative cells of adipose tissue for the treatment of post-irradiation vaginal-rectal fistula.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of radiation-induced rectovaginal fistula established at least six months after radiation therapy
* Absence of oncological disease relapse during whole observation period
* Absence of rectal and anal cancer
* Patient have read and signed informed consent

Exclusion Criteria:

* Contraindications for local/general anesthesia or a history of anesthetic medicines allergy
* Acute hemorrhoid or anal fissure
* Acute purulent paraproctitis
* Inflammatory colon diseases
* History of extensive posttraumatic or postoperative alterations which causes obstacles to follow protocol examination
* Chronic sub- or decompensated internal organs diseases
* Clinically significant laboratory tests abnormalities
* Conditions that limits patient compliance (dementia, psycho-neurological diseases, drug abuse, alcohol abuse etc.)
* Patients involved in other clinical trials or taking medications under research during last three months
* Cancer patients including postoperative chemo- or/and radiotherapy at least three months after surgery
* Patients with increased activated partial thromboplastin time level 1,8 times above normal
* Patients who take anticoagulants or took anticoagulants at least one month before including into trial
* Patients who take or took before investigation glycoprotein inhibitors IIB/IIIA
* Patients with history of taking medications that influence fatty tissue structure

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Serious adverse events | 4 weeks after injection of adipose-derived regenerative cells
  Frequency, type and severity of serious adverse events (SAE)
Serious adverse reactions | 4 weeks after injection of adipose-derived regenerative cells
  Frequency, type and severity of serious adverse reactions (SAR)

SECONDARY OUTCOMES:
Changes of fistula size | 48 weeks after intervention
  Intervention impact on dimensions of rectovaginal fistula
Changes in rectovaginal soft tissue density and flexibility | 48 weeks after intervention
  Intervention impact on soft tissue density and flexibility assessed by ultrasound elastography
Quality of life monitoring - 1 | 48 weeks after intervention
  Quality of life estimated by validated questionnaire: The Short Form (36) Health Survey (SF-36). SF-36 is a 36-item, patient-reported survey of patient health.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are:
  * vitality
  * physical functioning
  * bodily pain
  * general health perceptions
  * physical role functioning
  * emotional role functioning
  * social role functioning
  * mental health
Quality of life monitoring - 2 | 48 weeks after intervention
  Quality of life estimated by validated questionnaire. European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C-30 with module for proctitis-23 is a questionnaire developed to assess the proctitis-specific quality of life of cancer patients. Each subscale values varies from 1 to 4. Lower values represents better life quality. Total score is computed by summarizing of subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Georgy Dimov, PhD, Study Chair — South Ural State Medical University; Viacheslav Vasilyev, PhD, Study Director — South Ural State Medical University; Zhanna Teryushkova, PhD, Principal Investigator — South Ural State Medical University
Locations (1):
- South Ural State Medical University, Chelyabinsk, Chelyabinsk Oblast, Russia